CLINICAL TRIAL: NCT01368211
Title: PRESS Pathogen Reduction Extended Storage Study PRESS (Pathogen Reduction Extended Storage Study) A Pilot Study of Mirasol Platelets Treated in Platelet Additive Solution in Thrombocytopenic Patients
Brief Title: Mirasol-Treated Platelets - (Pathogen Reduction Extended Storage Study)
Acronym: PRESS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Part 1 completed, part 2 not done due to slow enrollment
Sponsor: Terumo BCTbio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CTS-0063
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Thrombocytopenia
Keywords: Mirasol; Thrombocytopenic; Pathogen reduction; Platelets; Thromboelastography; CCI; Corrected Count Increment
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirasol first, then Reference (Active Comparator): This study arm will receive first a 2-4-day-old Mirasol-treated platelets transfusion and then a reference 2-4-day-old untreated platelets transfusion (Mirasol-Reference sequence).
  Interventions: Biological: 2-4-day-old Mirasol-treated Platelets Transfusion; Biological: 2-4-day-old Untreated Platelets Transfusion
- Reference first, then Mirasol (Active Comparator): This study arm will receive first a reference 2-4-day-old untreated platelets transfusion and then a 2-4-day-old Mirasol-treated platelets transfusion (Reference-Mirasol sequence).
  Interventions: Biological: 2-4-day-old Mirasol-treated Platelets Transfusion; Biological: 2-4-day-old Untreated Platelets Transfusion

INTERVENTIONS:
Biological: 2-4-day-old Mirasol-treated Platelets Transfusion — 2-4-day-old Mirasol-treated Platelets Units with:
  * Platelet yield between 2.4x10e11 and 4.5x10e11
  * Plasma carryover of >32%
  * Cell count > 800x103/µL
  Other Names: Mirasol; Pathogen Reduction; PRT
Biological: 2-4-day-old Untreated Platelets Transfusion — 2-4-day-old Untreated Platelets Units with:
  * Platelet yield between 2.4x10e11 and 4.5x10e11
  * Plasma carryover of >32%
  * Cell count > 800x103/µL

SUMMARY:
The PRESS trial is a single-center, two-part, randomized cross-over pilot study in Copenhagen that will evaluate 1) the safety and performance of Mirasol-treated and untreated platelet products stored for 2-4 days and for 7-days in Platelet Additive Solution (PAS) and 2) the correlation between the TEG® parameters and platelet count increments after platelet transfusions in thrombocytopenic subjects.

DETAILED DESCRIPTION:
1. To evaluate in thrombocytopenic subjects the efficacy and safety of platelets treated with Mirasol Pathogen Reduction Technology (PRT) in Platelet Additive Solution. The following safety and efficacy measures will be compared between Mirasol treated and untreated platelets stored for 2-4 days and stored for 7 days:

   * Thrombelastography (TEG®) parameters: reaction time R, alpha angle α and maximal amplitude (MA)
   * Platelet Count Increment and Corrected Count Increment
   * Time to next platelet transfusion
   * Incidence of transfusion related (serious) adverse events
   * Incidence and severity of bleedings
2. To evaluate the use of the TEG® parameters as a measure for platelet transfusion efficacy and to evaluate the correlation between the TEG® parameters and the platelet Corrected Count Increments after platelet transfusions in thrombocytopenic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age of 18 years or older.
* Have thrombocytopenia or expected to develop thrombocytopenia requiring at least 3 platelet transfusions.
* Woman of child bearing potential must have a negative serum or urine pregnancy test within 72 hours before randomization.
* Subjects must have signed and dated the Informed Consent Form before performing any protocol related procedure.

Exclusion Criteria:

* History of any hypersensitivity reaction to riboflavin or metabolites.
* History of refractoriness to platelet transfusions (defined as 2 successive CCI1hr<5000) or presence of human leukocyte antigen (HLA) antibodies or positive lymphocytotoxicity or previously documented alloimmunization.
* Previous exposure to PRT-treated platelet concentrates.
* Active bleeding requiring one or more red cells concentrate transfusions (i.e. grade 3 or 4 bleeding according to the WHO bleeding assessment scale in Appendix 1).
* Exposure to an investigational product, within 30 days before randomization.
* Splenomegaly (presence of a palpable spleen whose border could be felt more than 4 cm below the costal margin) or splenectomy.
* History or diagnosis of Immune/Idiopathic Thrombocytopenic Purpura (ITP), Thrombotic Thrombocytopenia Purpura (TTP), or Haemolytic Uremic Syndrome (HUS).
* Use of prohibited medication (see section 5.5).
* Pregnant or lactating females.
* Any medical condition or treatment that would be expected to compromise the effectiveness of a platelet transfusion or that would interfere with an expected platelet count increment.
* Any other medical condition that would compromise the participation of the subject in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pär Johansson, MD, Principal Investigator — Transfusion Service Rigshospitalet - Dept of Immunology, Copenhagen Denmark; Lene Udby, MD, Principal Investigator — Hematology Service Rigshospitalet, Copenhagen Denmark
Locations (1):
- Hematology Service Rigshospitalet, Copenhagen, Blegdamsvej, Denmark

REFERENCES:
- [Result] Johansson PI, Simonsen AC, Brown PN, Ostrowski SR, Deberdt L, Van Hoydonck P, Yonemura SS, Goodrich RP. A pilot study to assess the hemostatic function of pathogen-reduced platelets in patients with thrombocytopenia. Transfusion. 2013 Sep;53(9):2043-52. doi: 10.1111/trf.12055. Epub 2012 Dec 24. PMID 23278371

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 patients enrolled versus 15 patients started: One patient was enrolled by error (exclusion criteria) and excluded after randomization.
Groups:
- Mirasol First, Then Reference: This study arm received first a Mirasol treated 2-4-day-old platelet transfusion and then a reference 2-4-day-old platelet transfusion (Mirasol-Reference sequence).
  Mirasol-treated Platelets: Mirasol-treated platelet units with:
  * Platelet yield between 2.4x10e11 and 4.5x10e11
  * Plasma carryover of >32%
  * Cell count > 800x103/µL
- Reference First, Then Mirasol: This study arm received first a reference untreated 2-4-day-old platelet transfusion and then a Mirasol treated 2-4-day-old platelet transfusion (Reference-Mirasol sequence).
  Mirasol-treated Platelets: Mirasol-treated platelet units with:
  * Platelet yield between 2.4x10e11 and 4.5x10e11
  * Plasma carryover of >32%
  * Cell count > 800x103/µL
Period: First Platelets Transfusion
Arm/Group | Mirasol First, Then Reference | Reference First, Then Mirasol
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Platelets Transfusion
Arm/Group | Mirasol First, Then Reference | Reference First, Then Mirasol
Started | 8 | 7
Completed | 7 | 5
Not Completed | 1 | 2
Not completed — No need for additional transfusion | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Mirasol First, Then Reference: This study arm will receive first a Mirasol treated 2-4-day-old platelet transfusion and then a reference 2-4-day-old platelet transfusion (Mirasol-Reference sequence).
  Mirasol-treated Platelets: Mirasol-treated platelet units with:
  * Platelet yield between 2.4x10e11 and 4.5x10e11
  * Plasma carryover of >32%
  * Cell count > 800x103/µL
- Reference First, Then Mirasol: This study arm will receive first a reference untreated 2-4-day-old platelet transfusion and then a Mirasol treated 2-4-day-old platelet transfusion (Reference-Mirasol sequence).
  Mirasol-treated Platelets: Mirasol-treated platelet units with:
  * Platelet yield between 2.4x10e11 and 4.5x10e11
  * Plasma carryover of >32%
  * Cell count > 800x103/µL
- Total: Total of all reporting groups
Arm/Group | Mirasol First, Then Reference | Reference First, Then Mirasol | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.13 (12.76) | 55.29 (19.95) | 57.33 (15.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  Denmark | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Amplitude at 1-hour Post-transfusion
Description: Thromboelastography (TEG) Parameter: Pre- to post-transfusional modification of Maximum Amplitude at 1-hour post-transfusion
Time Frame: pre-transfusion, 1-hour post transfusion
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Mirasol: Mirasol-treated 2-4-day old platelet transfusion
- Untreated Reference: Untreated 2-4-day old platelet transfusion
Arm/Group | Mirasol | Untreated Reference
Number analyzed (Participants) | 9 | 9
mm | 9.4 (7.0) | 15.4 (6.1)

2. Secondary Outcome: Change in Maximum Amplitude at 24-hours Post-transfusion
Description: Thromboelastography parameter: Pre- to post-transfusional modification in Maximum Amplitude at 24-hours post-transfusion
Time Frame: pre-transfusion, 24-hour post transfusion
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Mirasol | Untreated Reference
Number analyzed (Participants) | 9 | 9
mm | 10.4 (8.0) | 8.4 (4.7)

ADVERSE EVENTS:
Time Frame: 24 hours from start of transfusion
Description: Only transfusion related events
Groups:
- Mirasol-treated Platelets: Patients that received a Mirasol treated 2-4-day-old platelet transfusion.
- Untreated Reference Platelets: Patients that received an untreated reference2-4-day-old platelet transfusion.
Arm/Group | Mirasol-treated Platelets | Untreated Reference Platelets
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
Small numbers of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less